CLINICAL TRIAL: NCT01423344
Title: Assessment of the Value of the Free Kappa and Free Lambda Light Chain Assay in Clinical Evaluation of Response to Treatment
Brief Title: Clinical Evaluation of the Serum Free Light Chain Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charlotte Toftmann Hansen (Other)
Responsible Party: Sponsor-Investigator, Charlotte Toftmann Hansen, Fellow, ph.d-stud, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Other Study IDs: HFE-05-02; Danish Ethics comittee (Other: S-VF-20050035)
Record Dates: First submitted 2011-08-24; First posted 2011-08-25 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Free light chains
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: in patients with multiple myeloma there is a raised level of a protein, named M-protein. This M-protein is normally used to monitor disease status and evaluate response to treatment, as a decrease in M-protein is taken as evidence of therapeutic efficacy. However, the M-protein has a long half life in serum, approximately three weeks, which tend to be a practical problem, since the investigators can first determine hereafter if the treatment is effective.

A new assay has the possibility only to measure part of this protein, namely "the light chains", which also is measured in a blood sample. The half life of these light chains is much shorter, namely 2-6 hours. In theory, this means a more rapid measure of the effect of a given treatment, thereby being able to determine earlier if the treatment should continue or changed to another strategy.

Purpose: the purpose of this study is to evaluate the clinical value of the use of the serum free light chain (sFLC) assay in comparison to the M-protein in monitoring patients under treatment for multiple myeloma.

Method: the investigators measure sFLC in patients receiving there 1st treatment, either at the time of diagnosis or in the relapse setting. sFLC is measured on a regular basis, and the results are compared to the M-protein.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple myeloma
* abnormal serum free light chains
* medical needs of anti-myeloma therapy
* receiving standard anti-myeloma therapy

Exclusion Criteria:

* dialysis
* normal serum free light chains
* dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed patients with multiple myeloma, with medical needs and known patients with multiple myeloma at there 1st relapse and medical needs
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Time to 50% reduction in the concentration of the abnormal serum free light chain compared to 50% reduction in M-protein | 1, 2, 3, 4 and 5 days, 2, 3 and 6 weeks after therapy,

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte T Hansen, Fellow, Principal Investigator — Department of Haematology, research unit
Locations (1):
- Department of Haematology, research unit, Odense C, Denmark